CLINICAL TRIAL: NCT00801801
Title: Pilot Phase IIa Study of Metronomic Chemotherapy With Taxotere (Docetaxel) Plus Nexavar (Sorafenib) as First-Line Therapy in Performance Status-2 Patients With Advanced Non-Squamous Cell Non-Small Cell Lung Cancer
Brief Title: Study of Low Dose Chemotherapy Plus Sorafenib as Initial Therapy for Patients With Advanced Non-Squamous Cell NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsors withdrew funding; preliminary efficacy data was not encouraging.
Sponsor: Francisco Robert,MD (Other)
Collaborators: Sanofi (Industry); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Francisco Robert,MD, Principal Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F080703006; UAB 0750 (Other: Institutional study protocol number)
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Results first posted 2013-06-19 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Non Squamous Cell Lung Cancer; Non Small Cell Lung Cancer
Keywords: Docetaxel; Sorafenib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metronomic Docetaxel + Sorafenib (Experimental): Subjects with advanced non-squamous cell non-small cell lung cancer with poor performance status will receive treatment in this non-randomized, open-label Phase II Study of Metronomic Chemotherapy (docetaxel) plus sorafenib as first-line therapy.
  Subjects will be treated with metronomic chemotherapy with low dose docetaxel weekly for 3 out of 4 weeks, and sorafenib will be administered continuously 400 mg bid on a 28 day cycle. Treatment with metronomic chemotherapy will be expressed as a 4-week cycle.
  Interventions: Drug: Docetaxel + Sorafenib

INTERVENTIONS:
Drug: Docetaxel + Sorafenib — Subjects will be treated with metronomic chemotherapy with low dose docetaxel weekly for 3 out of 4 weeks, and sorafenib will be administered continuously 400 mg bid on a 28 day cycle. Treatment with metronomic chemotherapy will be expressed as a 4-week cycle. Tumor response to treatment will be evaluated after every 8 weeks. Treatment with metronomic chemotherapy and sorafenib will continue for a total of 6 cycles unless there is evidence of disease progression, intolerable toxicity, or withdrawal of consent. Maintenance therapy with sorafenib will then continue until disease progression, intolerable toxicity or withdrawal of consent.
  Other Names: Taxotere (Docetaxel); Nexavar (Sorafenib)

SUMMARY:
The purpose of this study is to assess the 2-month progression-free survival in patients with advanced or metastatic, non-squamous cell lung cancer treated with weekly low dose docetaxel in combination with a biologic dose of sorafenib.

DETAILED DESCRIPTION:
The median survival of untreated advanced stage NSCLC is 5-6 months (2,3). Patients with poor performance status due to malignancy or co-morbidities have a poorer survival. This group of patients is underrepresented in clinical trials and may not receive chemotherapy due to fear of increased toxicities with systemic chemotherapy. The overall median survival of patients with advanced NSCLC treated with first-line platinum-based doublets is less than 12 months (8 10 months) with a 1-year and 2-year survival rate of 33% and 11%, respectively (4 6). No chemotherapy regimen has a significant advantage over the others in the treatment of advanced NSCLC. Agents targeting epidermal growth factor receptor, matrix metalloproteinase, farnesyl transferase, protein kinase C and retinoic X receptor have so far shown no survival benefit in combination with chemotherapy in advanced NSCLC (7-13). Docetaxel has activity in NSCLC in both first line and second line settings. In poor performance status patients or elderly patients, single agent chemotherapy is recommended. Weekly docetaxel administration is well tolerated and has lesser incidence of hematologic toxicity with no difference in overall survival when compared to patients receiving higher doses (75 mg/m2) q 3 weeks (14-18). There is an increased need for better strategies to improve survival as well as reduce regimen related toxicity for this large group of patients. The use of targeted therapy as well as low dose-protracted chemotherapy (metronomic chemotherapy) needs evaluation as such therapies have a better toxicity profile.

Sorafenib (BAY 49-bursts of toxic maximum tolerated dose (MTD) chemotherapy interspersed with long breaks, there is now a shift in thinking towards the view that more compressed or accelerated schedules of drug administration using much smaller individual doses than the MTD would be more effective; not only in terms of reducing certain toxicities, but perhaps even in improving antitumor effect as well. Moreover, some of these dosing/scheduling strategies are ideally suited to combining chemotherapeutic agents with many of the new targeted biologic drugs. The most recent refinement of this concept is called "metronomic" chemotherapy, which refers to the frequent administration of cytotoxic chemotherapeutic agents at doses significantly below the MTD, with no prolonged drug-free breaks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic-proven non-squamous cell-NSCLC
* Advanced non-squamous-NSCLC: Stage IIIB with pleural effusion or stage IV, or recurrent disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status 2: In bed less than 50% of the time, unable to work, but able to care for self
* Measurable or non-measurable disease as defined by solid tumor response criteria (RECIST)
* No prior systemic chemotherapy or biologic therapy
* Age greater than or equal to 19 years old (Note: State of Alabama requirement)
* Adequate bone marrow and renal function as assessed by the following:

  * Hemoglobin greater than or equal to 9.0 g/dL
  * Absolute neutrophil count (ANC)greater than or equal to 1500/mm3
  * Platelet count greater than or equal to 100,000/mm3
  * Creatinine less than or equal to 1.5 times upper limit of normal (ULN)
* Hepatic function requirements

  * Total bilirubin less than or equal to ULN
  * AST and ALT and alkaline phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the two values (AST and ALT) should be used
* Women of childbearing potential must have a negative serum pregnancy test performed within 72 hours prior to the start of treatment.

Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation.

Men should use adequate birth control for at least three months after the last administration of sorafenib.

* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study-specific procedures.
* International normalized ratio (INR) less than or equal to 1.5 or a prothrombin time/partial prothrombin time (PT/PTT) within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.

Exclusion Criteria:

* Predominant squamous cell histology will be excluded
* Cardiac disease: Congestive heart failure greater than class II New York Heart Association (NYHA). Patents must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic pressure greater than 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 2.
* Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* History of significant hemoptysis (defined as bright red blood of a ½ teaspoon or more). Patients with blood-tinged or blood-streaked sputum will be permitted on study if the hemoptysis amount to less than 5 mL of blood per episode and less than 10 mL of blood per 24 hour period.
* Any other hemorrhage/bleeding event greater than or equal to CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.
* History of severe hypersensitivity reaction to any drugs formulated with polysorbate 80.
* Women who are breast-feeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: January 2008, Primary Completion Date: October 2009 and Study Completion Date: March 2011. Recruitment location: University of Alabama at Birmingham.
Pre-assignment Details: This study is to evaluate the use of targeted therapy as well as low dose-protracted chemotherapy (metronomic chemotherapy) in patients with advanced or metastatic non-squamous cell lung cancer (NSCLC). There is an increased need for better strategies to improve survival as well as reduce regimen related toxicities for this large group of patients.
Groups:
- Metronomic Taxotere and Nexavar: Subjects with advanced non-squamous cell non-small cell lung cancer with poor performance status will receive treatment in this non-randomized, open-label Phase II Study of Metronomic Chemotherapy (docetaxel) plus sorafenib as first-line therapy.
  Subjects will be treated with metronomic chemotherapy with low dose docetaxel weekly for 3 out of 4 weeks, and sorafenib will be administered continuously 400 mg bid on a 28 day cycle. Treatment with metronomic chemotherapy will be expressed as a 4-week cycle. Tumor response to treatment will be evaluated after every 8 weeks. Treatment with metronomic chemotherapy and sorafenib will continue for a total of 6 cycles unless there is evidence of disease progression, intolerable toxicity, or withdrawal of consent. Maintenance therapy with sorafenib will then continue until disease progression, intolerable toxicity or withdrawal of consent.
Period: Overall Study
Arm/Group | Metronomic Taxotere and Nexavar
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects with advanced non-squamous cell non-small cell lung cancer with poor performance status will receive treatment in this non-randomized, open-label Phase II Study of Metronomic Chemotherapy (docetaxel) plus sorafenib as first-line therapy.
Groups:
- Metronomic Taxotere + Nexavar: Subjects with advanced non-squamous cell non-small cell lung cancer with poor performance status will receive treatment in this non-randomized, open-label Phase II Study of Metronomic Chemotherapy (docetaxel) plus sorafenib as first-line therapy.
Arm/Group | Metronomic Taxotere + Nexavar
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: 2-month Progression-free Survival Rate
Description: Evaluation of the 2-month progression-free survival in poor performance status patients with non-squamous non-small cell lung cancer with the goal to improve 2-month progression free survival from 50% to 70%. The 2-month progression free survival is determined after 8 weeks on treatment. Those patients that had less than 20% increase in the tumor target lesions are considered as progression free survival. The primary endpoint is the percentage of patients that are progression free in 2 months.
Time Frame: Baseline to 2 months
Population: As the study did not accrue the maximum sample size for statistical analysis, none were done.
Measure: Number; unit: participants
Arm/Group | Metronomic Taxotere + Nexavar
Number analyzed (Participants) | 5
participants | 4

2. Secondary Outcome: Response Rate in Poor Performance Status Subjects
Description: To assess response rate and tumor control rate (complete remission + partial remission + stable disease) in poor performance status (PS =2) patients with advanced or metastatic (Stage IIIB - pleural effusion/IV) non-squamous cell-NSCLC treated with metronomic chemotherapy plus sorafenib. The objective response was defined as a percentage of those patients that had 30% or more of tumor regression at any time during treatment. Tumor control rate include the percentage of those patients that have less than 20% increase in the target tumor parameters during treatment (stable disease + partial response + complete response).
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Metronomic Docetaxel + Sorafenib
Number analyzed (Participants) | 5
participants | 0

ADVERSE EVENTS:
Time Frame: Toxicity assessment was performed on a weekly up to 6 months.
Groups:
- Metronomic Taxotere and Nexavar: Subjects with advanced non-squamous cell non-small cell lung cancer with poor performance status will receive treatment in this non-randomized, open-label Phase II Study of Metronomic Chemotherapy (docetaxel) plus sorafenib as first-line therapy.
Arm/Group | Metronomic Taxotere and Nexavar
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronomic Taxotere and Nexavar (N=5)
Pulmonary Embolism (Cardiac disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronomic Taxotere and Nexavar (N=5)
Fatigue (General disorders) | 2 (2)
Nausea & Vomiting (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hyperbilirubenemia (Hepatobiliary disorders) | 1 (1)
Transaminases (Hepatobiliary disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study initially sought to accrue a maximum sample size of 43 subjects. However, due to subjects' measured response and levels of clinical benefit in addition to a cut in funding, the study was stopped early and terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No